CLINICAL TRIAL: NCT06699680
Title: A Phase 1, Randomized, Double-Blind, Sponsor-Open, Placebo Controlled, First in Human Study to Evaluate the Safety, Tolerability, Immunogenicity, and Pharmacokinetics of Single Ascending and Multiple Doses of PRX019 in Healthy Adults
Brief Title: Phase 1 Study of PRX019 in Healthy Adult Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Prothena Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRX019-101
Record Dates: First submitted 2024-10-28; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants Study

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRX019, single dose (Experimental): Specified dose on specified days
  Interventions: Drug: PRX019; Drug: Placebo
- PRX019, multiple dose (Experimental): Specified dose on specified days
  Interventions: Drug: PRX019; Drug: Placebo

INTERVENTIONS:
Drug: PRX019 — Specified dose on specified days
Drug: Placebo — Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of PRX019 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are healthy as determined by the investigator based on review of medical history, physical examination, and clinical laboratory tests obtained during the screening period
* Participant is willing and able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, or clinical laboratory tests beyond what is consistent with a healthy population in the region in which the study is conducted
* Participant was exposed to an investigational drug (new chemical entity) within 90 days preceding the first dose administration, or within 7 times the elimination half-life, if known (whichever is longer)

NOTE: Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 6 months
Number of participants with clinical laboratory assessment abnormalities | Up to 6 months

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 6 months
Time to the maximum measured plasma concentration (Tmax) | Up to 6 months
Area under the concentration-time curve from time 0 through the intended dosing interval (AUCͳ) | Up to 6 months
Terminal elimination half-life in plasma (t1/2) | Up to 6 months
Maximum observed plasma concentration at steady state (Cmax,ss) | Up to 6 months
Area under the concentration-time curve from time 0 through the intended dosing interval at steady state (AUCͳ,ss) | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chad Swanson, Study Director — Prothena Biosciences
Locations (1):
- Local Institution, Los Alamitos, California, United States

IPD SHARING:
Plan to Share IPD: No
Prothena will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.